CLINICAL TRIAL: NCT03184428
Title: Retro- and Prospective Monocentric Study to Evaluate the Rate of Posterior Capsule Opacification Following Cataract Surgery With Implantation of the MICS (Micro Incision Cataract Surgery) -IOL (Intraocular Lens) L313
Brief Title: Posterior Capsule Opacification Following Cataract Surgery With Implantation of the MICS IOL L313
Status: Completed | Type: Observational
Sponsor: Dietrich-Bonhoeffer-Klinikum (Industry)
Responsible Party: Sponsor
Other Study IDs: STN 05/15
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Posterior Capsule Opacification
Keywords: YAG-Laser Capsulotomy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Implantation of IOL L313: Patients who have undergone a cataract surgery with implantation of the monofocal MICS IOL L313 more than 3 Years ago will be asked about the Treatment for Postoperative observation and survey.
  Interventions: Other: Postoperative observation and survey

INTERVENTIONS:
Other: Postoperative observation and survey — For postoperative Observation with a survey we ask the patients (or in case of no information the ophthalmologist) whether they had undergone a YAG-Laser-Capsulotomy after Cataract-Surgery or not.

SUMMARY:
This study collects intra- and postoperative data from the patients´charts retrospectively and evaluates retro- and prospectively the rate of posterior capsule opacification (PCO) following implantation of the intraocular lens L 313.

DETAILED DESCRIPTION:
This study is a postmarket study without interventions. Within the Standard Care Cataract surgery the participants have been implanted with the intraocular lens L313 in the period between September 2009 and December 2013. As criterium for the PCO was considered the Nd:YAG capsulotomy.

In the first step of the study, data was collected from the patients´charts.

In the second phase, a questionaire was sent to the patients with no recent examination, asking them to answer whether or not participants received a laser procedure due to PCO. In doubt the participants could answer: "I am not certain". For this step the investigator ensured the positive Votum of the Ethic Committee of the University of Greifswald, Germany.

On the third step of the study, the patients that were not certain of having such a laser procedure or did not answer per post, will be contacted on telephone. By uncertainty or no answer on the telephone the family eye doctor will be contacted to receive the necessary information. If the eye doctor has lost contact to the patient, then this patient will be documented as lost-to-follow-up.

Excluded were the patients that live >50km from the Department of Ophthalmology in Neubrandenburg, as well as patients with intraoperative capsule tear.

For the statistical analysis was used the program STATISTICA (StatSoft, Hamburg, Germany) and the survival analysis using the Kaplan-Meier formula, the statistical significance using the Chi-squared test and Spearman-Rank corelation and the Bonferroni adjustment if the test was repeated.

The investigators compared these results with the results of other publication. In order to do that the investigators calculated the capsulotomy quote from this study according to the time of the PCO recorded on the other studies. Included were only comparing studies that also used YAG-capsulotomy as criterium for the PCO.

Furthermore secondary data was collected: age, gender, cutting length, core hardness, duration of whole operation, time of phaco-emulsification, phaco-energy, phaco-machine, combination with other operation, surgeon, power of IOL. This data will be taken in concern for the validity of this study.

ELIGIBILITY:
Inclusion Criteria:

* retrospective: Patients who have undergone a Cataract surgery with Implantation of IOL L313
* prospective: signed informed consent

Exclusion Criteria:

* capsule rupture
* patients with too much travel distance between study center and home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3785 (5549 eyes)
Sampling Method: Probability Sample
Enrollment: 3785 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Hoeh, Prof. Dr., Principal Investigator — Department of Ophthalmology, Neubrandenburg, Germany; Christoforos Stylianides, Study Chair — Department of Ophthalmology, Neubrandenburg, Germany
Locations (1):
- Dietrich-Bonhoeffer-Klinikum, Neubrandenburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Yes
results will be published in ophthalmological journals

REFERENCES:
- [Background] Apple DJ, Peng Q, Visessook N, Werner L, Pandey SK, Escobar-Gomez M, Ram J, Auffarth GU. Eradication of posterior capsule opacification: documentation of a marked decrease in Nd:YAG laser posterior capsulotomy rates noted in an analysis of 5416 pseudophakic human eyes obtained postmortem. Ophthalmology. 2001 Mar;108(3):505-18. doi: 10.1016/s0161-6420(00)00589-3. PMID 11237905
- [Background] Apple DJ, Peng Q, Visessook N, Werner L, Pandey SK, Escobar-Gomez M, Ram J, Whiteside SB, Schoderbeck R, Ready EL, Guindi A. Surgical prevention of posterior capsule opacification. Part 1: Progress in eliminating this complication of cataract surgery. J Cataract Refract Surg. 2000 Feb;26(2):180-7. doi: 10.1016/s0886-3350(99)00353-3. PMID 10683785
- [Background] Auffarth GU, Brezin A, Caporossi A, Lafuma A, Mendicute J, Berdeaux G, Smith AF; European PCO Study Group. Comparison of Nd : YAG capsulotomy rates following phacoemulsification with implantation of PMMA, silicone, or acrylic intra-ocular lenses in four European countries. Ophthalmic Epidemiol. 2004 Oct;11(4):319-29. doi: 10.1080/09286580490515116. PMID 15512993
- [Background] Chitkara DK, Smerdon DL. Risk factors, complications, and results in extracapsular cataract extraction. J Cataract Refract Surg. 1997 May;23(4):570-4. doi: 10.1016/s0886-3350(97)80216-7. PMID 9209994
- [Background] Meacock WR, Spalton DJ, Boyce JF, Jose RM. Effect of optic size on posterior capsule opacification: 5.5 mm versus 6.0 mm AcrySof intraocular lenses. J Cataract Refract Surg. 2001 Aug;27(8):1194-8. doi: 10.1016/s0886-3350(01)00855-0. PMID 11524189
- [Background] Menapace R. [After-cataract following intraocular lens implantation. Part II: prevention with alternative implants and techniques]. Ophthalmologe. 2007 Apr;104(4):345-53; quiz 354-5. doi: 10.1007/s00347-007-1505-1. German. PMID 17372739
- [Background] Menapace R. [After-cataract following intraocular lens implantation. Part I. Genesis and prevention by optimizing conventional lens implants and surgical techniques]. Ophthalmologe. 2007 Mar;104(3):253-62; quiz 263-4. doi: 10.1007/s00347-007-1492-2. German. PMID 17323043
- [Background] Mester U, Fabian E, Gerl R, Hunold W, Hutz W, Strobel J, Hoyer H, Kohnen T. Posterior capsule opacification after implantation of CeeOn Edge 911A, PhacoFlex SI-40NB, and AcrySof MA60BM lenses: one-year results of an intraindividual comparison multicenter study. J Cataract Refract Surg. 2004 May;30(5):978-85. doi: 10.1016/j.jcrs.2003.09.052. PMID 15130632
- [Background] Nishi Y, Ikeda T, Nishi K, Mimura O. Epidemiological evaluation of YAG capsulotomy incidence for posterior capsule opacification in various intraocular lenses in Japanese eyes. Clin Ophthalmol. 2015 Sep 1;9:1613-7. doi: 10.2147/OPTH.S89966. eCollection 2015. PMID 26366054
- [Background] Pandey SK, Apple DJ, Werner L, Maloof AJ, Milverton EJ. Posterior capsule opacification: a review of the aetiopathogenesis, experimental and clinical studies and factors for prevention. Indian J Ophthalmol. 2004 Jun;52(2):99-112. PMID 15283214
- [Background] Prosdocimo G, Tassinari G, Sala M, Di Biase A, Toschi PG, Gismondi M, Corbanese U. Posterior capsule opacification after phacoemulsification: silicone CeeOn Edge versus acrylate AcrySof intraocular lens. J Cataract Refract Surg. 2003 Aug;29(8):1551-5. doi: 10.1016/s0886-3350(02)02051-5. PMID 12954304
- [Background] Schaumberg DA, Dana MR, Christen WG, Glynn RJ. A systematic overview of the incidence of posterior capsule opacification. Ophthalmology. 1998 Jul;105(7):1213-21. doi: 10.1016/S0161-6420(98)97023-3. PMID 9663224
- [Background] Schmidbauer JM, Vargas LG, Apple DJ, Auffarth GU, Peng Q, Arthur SN, Escobar-Gomez M. [Millenniums update on posterior capsule opacification (PCO) scores, centration, biocompatibility and fixation of foldable intraocular lenses (IOL) - an analysis of 1,221 pseudophakic post mortem globes]. Klin Monbl Augenheilkd. 2001 Oct;218(10):649-57. doi: 10.1055/s-2001-18386. German. PMID 11706380
- [Background] Schriefl SM, Leydolt C, Stifter E, Menapace R. Posterior capsular opacification and Nd:YAG capsulotomy rates with the iMics Y-60H and Micro AY intra-ocular lenses: 3-year results of a randomized clinical trial. Acta Ophthalmol. 2015 Jun;93(4):342-7. doi: 10.1111/aos.12543. Epub 2014 Nov 13. PMID 25393894
- [Background] Spyridaki M, Hoh H. [Comparison of four MICS intraocular lenses regarding their rates of neodymium:YAG laser capsulotomy]. Klin Monbl Augenheilkd. 2010 Mar;227(3):208-14. doi: 10.1055/s-0028-1109853. Epub 2010 Mar 16. German. PMID 20234985
- [Background] Tetz MR, Nimsgern C. Posterior capsule opacification. Part 2: Clinical findings. J Cataract Refract Surg. 1999 Dec;25(12):1662-74. doi: 10.1016/s0886-3350(99)00259-x. PMID 10609214
- [Background] Wehner W. [Microincision intraocular lens with plate haptic design. Evaluation of rotational stability and centering of a microincision intraocular lens with plate haptic design in 12-19 months of follow-up]. Ophthalmologe. 2007 May;104(5):393-4, 396-8. doi: 10.1007/s00347-007-1500-6. German. PMID 17384950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eyes of patients who underwent a cataract surgery in the Department of Ophthalmology in Neubrandenburg between September 2009 and December 2013 and had an L313 MICS lens implanted.
Pre-assignment Details: The following reasons led to an exclusion of participants:
  * intraoperative posterior capsule rupture
  * Distance between place of residence and place of investigation >50 km
  * Exchange of the intraocular lens
  * Practice closure of the supervising ophthalmologist
  * no entry in any established doctor's medical system
  * no follow-up
Units Other Than Participants: eyes
Groups:
- L313-Implantation: Eyes of patients who underwent a cataract surgery in the Department of Ophthalmology in Neubrandenburg between September 2009 and December 2013 and had an L313 MICS lens.
Period: Overall Study
Arm/Group | L313-Implantation
Started | 3785; 5549 eyes
Completed | 2963; 4388 eyes
Not Completed | 822; 1161 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Implantation of IOL L313: Patients who have undergone a cataract surgery with implantation of the monofocal MICS IOL L313 more than 3 Years ago will be asked about the treatment for postoperative observation and survey.
  Postoperative observation and survey: For postoperative observation with a survey we ask the patients (or in case of no information the ophthalmologist) whether they had undergone a Nd: YAG-Laser-Capsulotomy after Cataract-Surgery or not.
Arm/Group | Implantation of IOL L313
Number analyzed (Participants) | 3785
Number analyzed (eyes) | 5549
Age, Categorical [Count of Units; unit: eyes]
  <=18 years | 2
  Between 18 and 65 years | 886
  >=65 years | 4661
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.75 (9.06)
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 3285
  Male | 2264
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Posterior Capsule Opacification Following Implantation of IOL 313 up to 8 Years
Description: In order to find out whether patients with cataract surgery are affected by lens opacification, we assessed whether a Nd:YAG laser capsulotomy was performed for treatment.
  For this purpose, the patient files were spotted first. Those who had no recent findings were asked in writing if and when a laser treatment was performed. In the absence of feedback and in case of uncertain or unusable written answer, a telephone consultation with the patient was made. If sufficient information was not available afterwards, the ophthalmologist was asked for information (by phone, by written request or by collecting the data on site in the practices).
Time Frame: up to 8 years
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Implantation of IOL L313 Age<55: Patients age<55 who have undergone a cataract surgery with implantation of the monofocal MICS IOL L313 more than 3 Years ago will be asked about the Treatment for Postoperative observation and survey.
- Implantation of IOL L313 Age≥55: Patients age≥55 who have undergone a cataract surgery with implantation of the monofocal MICS IOL L313 more than 3 Years ago will be asked about the Treatment for Postoperative observation and survey.
Arm/Group | Implantation of IOL L313 Age<55 | Implantation of IOL L313 Age≥55
Number analyzed (Participants) | 111 | 2852
Number analyzed (eyes) | 164 | 4224
percentage of eyes
  1 year | 7.9 | 4.7
  2 years | 17.1 | 8.2
  after 4 years | 25.0 | 17.2
  after 6 years | 25.6 | 22.4

2. Secondary Outcome: Correlation Coefficient Between Capsulotomy Rate and Parameters
Description: Correlation coefficients between capsulotomy rate and patient parameters:
  1. age
  2. gender,
     and surgical parameters:
  3. cutting length,
  4. core hardness,
  5. duration of whole operation,
  6. time of phaco-emulsification,
  7. phaco-energy,
  8. phaco-machine,
  9. combination with other operation,
  10. surgeon,
  11. power of IOL.
Time Frame: up to 8 years
Measure: Number; unit: Correlation coefficient
Units Other Than Participants: eyes
Groups:
- Capsulotomy Rate/Age: Correlation coefficient between capsulotomy rate and age
- Capsulotomy Rate/Gender: Correlation coefficient between capsulotomy rate and gender
- Capsulotomy Rate/Cutting Lenth: Correlation coefficient between capsulotomy rate and cutting length
- Capsulotomy Rate/Core Hardness: Correlation coefficient between capsulotomy rate and core hardness
- Capsulotomy Rate/Duration of Whole Operation: Correlation coefficient between capsulotomy rate and duration of whole operation
- Capsulotomy Rate/Time of Phaco-emulsification: Correlation coefficient between capsulotomy rate and time of phaco-emulsification
- Capsulotomy Rate/Phaco-energy: Correlation coefficient between capsulotomy rate and phaco-energy
- Capsulotomy Rate/Phaco-machine: Correlation coefficient between capsulotomy rate and phaco-machine
- Capsulotomy Rate/Combination With Other op: Correlation coefficient between capsulotomy rate and L-313 implantation in combination with other op
- Capsulotomy Rate/Surgeon: Correlation coefficient between capsulotomy rate and surgeon
- Correlation Rate/Power of IOL: Correlation coefficient between capsulotomy rate and power of IOL
Arm/Group | Capsulotomy Rate/Age | Capsulotomy Rate/Gender | Capsulotomy Rate/Cutting Lenth | Capsulotomy Rate/Core Hardness | Capsulotomy Rate/Duration of Whole Operation | Capsulotomy Rate/Time of Phaco-emulsification | Capsulotomy Rate/Phaco-energy | Capsulotomy Rate/Phaco-machine | Capsulotomy Rate/Combination With Other op | Capsulotomy Rate/Surgeon | Correlation Rate/Power of IOL
Number analyzed (Participants) | 2963 | 2852 | 2852 | 2929 | 3036 | 3017 | 2857 | 2990 | 2852 | 3784 | 2852
Number analyzed (eyes) | 4388 | 4224 | 4224 | 3944 | 4068 | 4088 | 3864 | 3906 | 4224 | 4049 | 4224
Correlation coefficient | 0.0001 | 0.276 | 0.578 | 0.041 | 0.467 | 0.739 | 0.782 | 0.746 | 0.002 | 0.727 | 0.578
Statistical Analysis 1: Comparison: Capsulotomy Rate/Age vs Capsulotomy Rate/Gender vs Capsulotomy Rate/Cutting Lenth vs Capsulotomy Rate/Core Hardness vs Capsulotomy Rate/Duration of Whole Operation vs Capsulotomy Rate/Time of Phaco-emulsification vs Capsulotomy Rate/Phaco-energy vs Capsulotomy Rate/Phaco-machine vs Capsulotomy Rate/Combination With Other op vs Capsulotomy Rate/Surgeon vs Correlation Rate/Power of IOL; Test type: Other; p < 0.05, Spearman's rank-order correlation; Bonferroni adjustment in addition

ADVERSE EVENTS:
Time Frame: n/a All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed because no interventions were performed in the Department of Ophthalmology (only a questionnaire for information sampling was required).
Description: No interventions were performed in the Department of Ophthalmology (only a questionnaire for information sampling was required), thus adverse events were not monitored (including Serious Adverse Events, All-Cause-Mortality, Other Adverse Events). An investigation would have been necessary only in case of low patient's response.
Arm/Group | Implantation of IOL L313
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03184428/Prot_SAP_000.pdf